CLINICAL TRIAL: NCT01657500
Title: A Randomized, Prospective, Double Masked Clinical Trial of Life 4°C Versus Optisol GS Corneal Storage Media
Brief Title: Life 4°C Versus Optisol in Corneal Storage Media
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Lass, M.D., Charles I Thomas Professor and Chairman CWRU Department of Ophthalmology and Visual Sciences Director, University Hospitals Eye Institute, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 11-10-20
Record Dates: First submitted 2012-07-17; First posted 2012-08-06 (Estimated); Results first posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Complications of Corneal Transplant
Keywords: endothelial keratoplasty
MeSH Terms: interventions — Chondroitin Sulfates; Dextrans; Gentamicins; Complex Mixtures; Culture Media, Serum-Free

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Life 4°C media for cornea storage (Active Comparator): Donor cornea is stored in the Life 4°C media prior to implantation.
  Interventions: Other: Life 4°C solution for cornea storage
- Optisol GS (Active Comparator): Donor cornea is stored in the Optisol GS media prior to implantation.
  Interventions: Other: Corneal donor storage in Optisol GS media solution

INTERVENTIONS:
Other: Corneal donor storage in Optisol GS media solution — Donor tissue is preserved in the Optisol media until ready for implantation
  Other Names: Chondroitin Sulfates; Dextrans; Gentamicins; Complex Mixtures; Culture Media, Serum Free
  Arms: Optisol GS
Other: Life 4°C solution for cornea storage — Donor cornea is stored in the Life 4°C media prior to implantation.
  Other Names: Chondroitin Sulfates; Dextrans; Gentamicins; Streptomicins; Complex Mixtures; Culture Media, Serum Free
  Arms: Life 4°C media for cornea storage

SUMMARY:
The purpose of this study is to compare the success of storing a donor cornea in Optisol GS, the current standard vs. storing the donor cornea in Life4°C, a newer solution. The donor cornea to be used for EK will be provided by an eye bank and will have been stored in either an Optisol GS solution or a Life 4°C solution. At 6 months, the doctors will determine whether there are any comparable differences in cell loss and graft clarity between the two donor corneas.

DETAILED DESCRIPTION:
1. Purpose/ Specific Aims

   The purpose of this study is to compare the success of storing a donor cornea in Optisol GS, the current standard solution that the donor cornea is stored in prior to surgery versus storing the donor cornea in Life 4°C, a newer solution. Laboratory tests that led to the recent approval of this new storage solution by the Food and Drug Administration have suggested that this solution may support the health of the endothelial cells better than Optisol GS. While there is extensive in vitro and ex vivo data regarding Life 4°C and its transport chamber, there are no short or long term in vivo studies to examine its performance clinically and the relationship of its performance to Optisol GS and its transport chamber. This study has been designed to examine these questions.

   1.1 STUDY OBJECTIVES Primary objective: To determine whether endothelial cell loss post EK is comparable 6 months postoperatively for donor corneas preserved in Life 4°C vs. Optisol GS corneal storage media

   Secondary objective: To determine whether graft clarity post EK is comparable 6 months postoperatively for donor corneas preserved in Life 4°C versus Optisol GS corneal storage media
2. Background and Significance

Currently it is estimated by the Eye Bank Association of America (EBAA) that 3500 to 5000 Americans wait an average of 1-2 months to undergo penetrating or endothelial keratoplasty. The situation worldwide is considerably more complex, and the availability of tissue is much more limited. In view of this shortage of tissue, much research has been undertaken with a view towards prolonging donor storage time and yet maintaining a viable endothelium, which is crucial to successful transplantation. Extended preservation time has transformed corneal transplantation surgery into an elective procedure and has facilitated the availability of available donor tissue. However, corneal preservation involves many other factors in addition to simply increasing the length of donor storage time.

The functional status of the endothelium, epithelium and sustained corneal deturgescence after corneal preservation are of great clinical importance and contribute primarily to the success of the surgical outcome. Other areas of concern to be addressed in the development of a complete corneal preservation medium include the enhancement of corneal wound healing and the reduction or elimination of the normal progressive loss of endothelial cells post keratoplasty. Preservation of existing endothelial cells during corneal preservation is important because endothelial cells continue to be lost after penetrating keratoplasty at a faster rate than normal aging1. Timely and adequate healing of corneal tissues is required to restore visual acuity.

The current "gold standard" in 4°C corneal preservation medium is Optisol GS (Bausch & Lomb Surgical, Inc.). This is an improved formulation of Optisol 2 (Chiron Vision, Irvine, CA, U.S.A.) modified by the addition of 200 µg/ml of streptomycin sulfate. Optisol preserved the corneal endothelium as well as DexSol (Chiron Vision, Irvine, CA, U.S.A.), the previous widely used corneal preservation medium, and was better at preventing stromal swelling during storage 2-5. The addition of streptomycin to gentamicin in corneal preservation media was effective against resistant strains of bacteria6. Optisol GS exhibited improved antibacterial activity without any increased toxicity to the endothelium7-8. In vitro studies of Optisol GS stored human corneas concluded that storage time at 4°C is limited by the inability to preserve corneal epithelium greater than 1 week, although 84% of the endothelium was deemed viable after three weeks of storage 9,10. A clinical study found that the probability of an epithelial defect 1 day after penetrating keratoplasty increased with increased storage time in Optisol GS11.

Optisol GS is a chondroitin sulfate containing medium supplemented with dextran, additional antioxidants, energy sources and nutritive substrates12. These components address the understanding that the cornea is still metabolically active at low storage temperatures. The composition of synthetic media must address the increased stromal hydration that occurs with increased preservation time and reduced temperatures. In the progression of intermediate-term corneal preservation medium development, dextran, an osmotic agent, was added in an effort to reduce the intraoperative rebound swelling associated with chondroitin sulfate containing medium. Chondroitin sulfate and dextran assist in the prevention of stromal hydration by increasing the colloidal osmotic pressure in the aqueous environment surrounding the stored cornea. Sustained corneal deturgescence during and after corneal preservation are of great clinical importance, reducing handling and suturing problems encountered by the transplant surgeon, thus reducing the risk of graft failure

A superior corneal preservation medium would maintain cellular viability while lengthening current storage times for more efficient use of donor tissue, prevent stromal swelling to facilitate keratoplasty, and eliminate or suppress microbiologic growth to prevent rare but catastrophic endophthalmitis.

2.1 INVESTIGATIONAL AGENT Life 4°C is an FDA approved, new advanced corneal preservation medium (30 ml) for storage of human corneas suitable for keratoplasty for up to 14 days under refrigeration (2-8°C). Life 4°C is sterile, non-pyrogenic, advanced buffered corneal preservation medium which is supplemented with chondroitin sulfate (membrane stabilizer), recombinant human insulin (cell metabolism enhancer), Dextran (osmotic agent), glutathione (antioxidant, free-radical scavenger, enzyme cofactor), stabilized L-glutamine, ATP precursors, nutrient cell supplements, amino acids, vitamins, trace elements, gentamycin, streptomycin and phenol red (pH indicator). Life 4°C has been formulated to be used to the full extent of corneal storage time, by preventing stromal swelling, maintaining corneal epithelium and providing optimum endothelial cell preservation.

In addition, TRANSEND is a new corneal storage, viewing and transport system. It was designed for performance to meet the challenges of extended storage, specular microscopy and shipping. TRANSEND viewing chamber is designed to accommodate larger scleral rims needed for the newest surgical procedures. The increased medium volume (30 ml) and greater fluid flow to the cornea reduces metabolic waste build-up, important to cellular health. Increased medium volume results in excellent corneal preservation with minimal corneal swelling during storage. The TRANSEND viewing chamber utilizes both a top seal and o-ring side seal for leak-proof performance. The cornea is held securely during storage, specular microscopy and shipping. The viewing chamber is gamma irradiated, therefore there are no ETO residuals. The use of new tamper seals eliminates the use of high temperature heat seals. The outer shipping container allows the inner viewing chamber to arrive dry and secure to the surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing EK for FECD only.
2. Age range of 30-85 years with minimum life expectancy of at least 1 year
3. Willingness to return to study site at 1 month, 3 months, and 6 months to complete study procedures
4. Permissible EK procedures with preoperative diagnoses

   * Pseudophakic FECD with posterior capsule supported or suture-fixated posterior chamber intraocular lens (IOL)
   * Phakic FECD
   * EK, phacoemulsification with posterior chamber IOL for phakic FECD with cataract
5. Stromal vascularization is acceptable
6. Controlled glaucoma on medication and/or previous trabeculectomy and laser trabeculoplasty is acceptable

Exclusion Criteria:

1. Since EK is suitable only for corneal conditions with endothelial dysfunction, all corneal conditions not associated with endothelial failure that are managed with PKP only are excluded (e.g. keratoconus, stromal dystrophies, traumatic corneal scars).

* Other exclusions include:
* Other primary endothelial dysfunction conditions including pseudophakic bullous keratopathy not due to FECD, posterior polymorphous corneal dystrophy and congenital hereditary corneal dystrophy
* Pseudophakic FECD with open loop anterior chamber IOL
* Previous failed keratoplasty, either EK or PKP
* Central subepithelial or stromal scarring detected preoperatively that could impact graft clarity assessment
* Anterior or peripheral anterior synechiae
* Uncontrolled glaucoma > 25 Hg with or without prior filtering surgery or shunt placement.
* Controlled glaucoma with tube shunt placement.
* Uncontrolled Uveitis - Fellow eye visual acuity < 20/200
* Fellow eye already included in the study

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lass, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (4):
- United States (4):
  - Price Vision Group, Indianapolis, Indiana
  - Verdier Eye Center, Grand Rapids, Michigan
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Central Pennsylvannia Eye Institute, Hershey, Pennsylvania

REFERENCES:
- [Derived] Price MO, Knight OJ, Benetz BA, Debanne SM, Verdier DD, Rosenwasser GO, Rosenwasser M, Price FW Jr, Lass JH. Randomized, prospective, single-masked clinical trial of endothelial keratoplasty performance with 2 donor cornea 4 degrees C storage solutions and associated chambers. Cornea. 2015 Mar;34(3):253-6. doi: 10.1097/ICO.0000000000000354. PMID 25625366

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Life 4°C Media for Cornea Storage | Optisol GS
Started | 32 | 32
Completed | 27 | 27
Not Completed | 5 | 5
Not completed — set impropperly matched | 3 | 3
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: age 30-85
Groups:
- Total: Total of all reporting groups
Arm/Group | Life 4°C Media for Cornea Storage | Optisol GS | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Customized [Number; unit: years]
  30-85 | 27 | 27 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Cell Loss Post EK for Donor Corneas Preserved in Life 4°C and Optisol GS Corneal Storage Media
Description: Endothelial cell loss and graft success were comparable at 6 months for paired donor corneas stored in Optisol GS and Life4°C.
Time Frame: Six months
Population: Male and female subjects aged from 30-85 years, had FECD, undergoing endothelial keratoplasty, Exclusion criteria: pseudophakic FECD with AC IOL, previous failed keratoplasty, synechiae, corneal scarring impacting graft clarity assessment, uncontrolled uveitis, fellow eye VA 20/200, uncontrolled glaucoma or having a tube shunt placement.
Measure: Mean (Standard Deviation); unit: % endothelial cell loss
Groups:
- Optisol GS: Time after keratoplasty Number of pairs Life 4°C (mean ± SD) Optisol GS (mean ± SD
Arm/Group | Optisol GS | Life 4C
Number analyzed (Participants) | 32 | 32
% endothelial cell loss | 20 (20) | 18 (18)
Statistical Analysis 1: Comparison: Optisol GS vs Life 4C; Main outcome measure was endothelial cell loss at 6 months after EK. Sample size and statistical power calculations for testing equivalence of means within 10% range were performed at 80% power/0.025 level of significance. 20% variability was assumed. 6-month endothelial cell loss) should not differ significantly for surgeon-prepared versus eye bank-prepared tissue. Assuming pairs of corneas matched by pt. diagnosis and other characteristics, the required sample size was 34 donor pairs; Test type: Non-Inferiority or Equivalence — See above; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Life 4°C Media for Cornea Storage: Donor cornea is stored in the Life 4°C media prior to transplantation.
  Life 4°C solution for cornea storage: Donor cornea is stored in the Life 4°C media prior to transplantation.
  Air was reinjected in 4 eyes to treat partial graft detachment. During the 6-month follow-up period, 1 graft experienced a graft rejection episode, which responded to increased topical corticosteroid therapy. 5 eyes had intraocular pressure (IOP) elevation requiring use of glaucoma medications or reduction of topicalcorticosteroid strength or dosing frequency. 2 eyes had laser capsulotomy to treat capsular haze. 1 eye had recurrent erosions because of peripheral bullae and was treated with lamellar keratectomy, and 1 eye was diagnosed with herpes simplex virus keratitis and was treated with antiviral medication. Altogether, 14 of 27 eyes (52%) in each corneal storage solution group had a postoperative intervention (P = 1.0).
- Optisol GS: Donor cornea is stored in the Optisol GS media prior to transplantation
  Corneal donor storage in Optisol GS media solution: Donor tissue is preserved in the Optisol media until ready for transplantation In the early postoperative period, 1 DSAEK graft in the Optisol GS group was repositioned because it fully detached. Air was reinjected in 2 eyes to treat partial graft detachment. During the 6-month follow-up period, 1 graft experienced a graft rejection episodes, which responded to increased topical corticosteroid therapy. 7 eyes had intraocular pressure (IOP) elevation requiring use of glaucoma medications or reduction of topical corticosteroid strength or dosing frequency. 2 eyes had laser capsulotomy to treat capsular haze. 1 eye had a vitreous strand associated with a capsular tear during cataract removal and was treated with laser vitreolysis.Altogether, 14 of 27 eyes (52%) in each corneal storage solution group had a postoperative intervention (P = 1.0).
Arm/Group | Life 4°C Media for Cornea Storage | Optisol GS
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes